CLINICAL TRIAL: NCT00047684
Title: Development and Initial Evaluation of Brief Integrative Therapy for PTSD
Brief Title: Brief Integrative Therapy for Post-Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21MH061319 (NIH); R21MH061319 (NIH); DSIR AT-AS
Record Dates: First submitted 2002-10-11; First posted 2002-10-16 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2008-09

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Child Abuse, Sexual
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Coitus

INTERVENTIONS:
Behavioral: Brief Integrative Therapy

SUMMARY:
The purpose of this study is to refine Brief Integrative Therapy (BIT) and to evaluate its effectiveness in treating women with Post-Traumatic Stress Disorder (PTSD) following childhood sexual abuse. This study will also promote the development of skills that are necessary for increasing quality of life and improving self-esteem.

DETAILED DESCRIPTION:
BIT integrates interpersonal, problem solving, affect regulation, and psychoeducational components. In this study, BIT is used to encourage women to focus on current issues and problems. The BIT therapist will help patients identify the impact of PTSD on their functioning, help them identify effective coping strategies for dealing with trauma-related distress, and encourage them to establish and maintain a certain degree of independence from the therapist.

Patients receive 15 weekly sessions of BIT. Assessments occur pre-treatment, post-treatment, and at a 3-month follow-up, and include self-report measures, clinician administered PTSD scale questions, interviews, and evaluations of lifetime stressors.

ELIGIBILITY:
Inclusion Criteria:

* Post-Traumatic Stress Disorder (PTSD) diagnosis
* Childhood sexual abuse, defined as any sexual contact before the age of 16 with someone 5 or more years older
* At least 1 clear, detailed memory of sexual abuse

Exclusion criteria:

* Substance abuse or dependence
* Psychotic disorder, bipolar disorder, or dissociative disorder
* 2 or more suicidal or parasuicidal acts in the past year
* Domestic violence involvement
* Pregnancy or attempting to become pregnant

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2001-11; Study Completion 2002-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for PTSD, White River Junction, Vermont, United States